CLINICAL TRIAL: NCT06945458
Title: A Phase 1b Open-label, Multicenter, Single-arm Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Clinical Activity of Orally Administered KT-621 in Adult Participants With Moderate to Severe Atopic Dermatitis
Brief Title: Safety, PK, PD, and Clinical Activity of Orally Administered KT-621 in Adult Patients With Atopic Dermatitis (AD)
Acronym: BroADen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kymera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KT621-AD-102
Record Dates: First submitted 2025-04-09; First posted 2025-04-25 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis
Keywords: KT621; STAT6; STAT6 degrader; Targeted protein degrader; Phase 1
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- KT-621 (Experimental): Each participant receives daily oral doses of KT-621 throughout the 28-day treatment period.
  Interventions: Drug: KT-621

INTERVENTIONS:
Drug: KT-621 — Oral drug

SUMMARY:
This is a study to evaluate safety, tolerability, pharmacokinetics, pharmacodynamics, and clinical activity of orally administered KT-621 in adult male and female patients with moderate to severe atopic dermatitis (AD).

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 18 to 55 years (inclusive) at the time of screening
* Participants must be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other procedures
* Participants must have had chronic atopic dermatitis (AD) for at least 1 year before Screening.
* Moderate to very severe eczema as determined by Eczema Area and Severity Index (EASI) score of at least 16 at the baseline visit.
* A validated Investigator Global Assessment (vIGA) score of at least 3 at the baseline visit, indicating moderate to severe AD.
* At least 10% body surface area (BSA) of AD involvement at the baseline visit.
* Weekly average Peak Pruritus Numeric Rating Scale (NRS) of at least 4 at the baseline visit.
* Documented history within 6 months prior to baseline visit of either inadequate response or contraindication to topical medications for AD.
* Application of stable dose of moisturizer at least twice daily for at least 7 consecutive days immediately prior to the baseline visit.

Exclusion Criteria:

* Participants who have a clinically relevant history of respiratory, gastrointestinal (GI), renal, hepatic, hematological, lymphatic, endocrinological, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, ophthalmological, or connective tissue diseases or disorders.
* Participants who have any surgical or medical procedure planned during participation in the study.
* Participants with a history of alcohol or substance abuse within the previous 2 years.
* Participants who have any known factor, condition, or disease that might interfere with treatment compliance, study conduct or interpretation of the results.
* Participants whose results from clinical laboratory safety tests are outside the local reference range at Screening.
* Participants who have been dosed with any investigational drug or device in a clinical study within 8 weeks or 5 half-lives (whichever is longer) of KT-621 administration.
* Participants with a history of lack of response to any medication targeting interleukin (IL)-4, IL-13, and/or janus kinase (JAK)- signal transducer and activator of transcription (STAT) pathways (e.g. dupilumab, tralokinumab, upadacitinib, abrocitinib) at approved doses after at least 16 weeks of therapy.
* Pregnant or breastfeeding women, or women planning to become pregnant or breastfeed during the study.
* Female participants of childbearing potential with a positive or undetermined pregnancy result at the Screening and baseline visits.
* Participants with a known sensitivity to any of the components of KT-621.
* Participants who are a member of the investigational team or his/her immediate family.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) | From enrollment through the safety follow-up visit on Day 43
Incidence of treatment-emergent potentially clinically-significant abnormalities in electrocardiogram (ECG) results, vital signs, or laboratory test results from the serum chemistry, hematology (with differential), chemistry, or coagulation panels. | From enrollment through the safety follow-up visit on Day 43

SECONDARY OUTCOMES:
Plasma PK parameter estimates of KT-621 derived from plasma concentration-time data | From baseline visit through the safety follow-up visit on Day 43
  Trough concentrations taken at each visit before dosing, post-dose concentrations taken after dosing at Days 1 and 15.

OTHER OUTCOMES:
KT-621 concentrations in skin | From baseline visit through the safety follow-up visit on Day 43
Change in Eczema Area and Severity Index (EASI) score | From screening through the safety follow-up visit on Day 43
Proportion of participants who achieve a validated Investigator Global Assessment (vIGA) score of 0 or 1 at scheduled clinic visits | From screening through the safety follow-up visit on Day 43
  On a scale of 0 to 4, 0 being no inflammatory signs of AD, 4 being severe inflammatory signs of AD
Change from baseline in the Peak Pruritus Numeric Rating Scale (NRS) score | From baseline visit through the safety follow-up visit on Day 43
  Percent change from baseline
Change from baseline in levels of signal transducer and activator of transcription 6 protein, in skin and in whole blood | From baseline visit through the safety follow-up visit on Day 43
Change from baseline in the serum levels of Th2 biomarkers such as thymus and activation-regulated chemokine (TARC) | From baseline visit through the safety follow-up visit on Day 43
Change from baseline through Week 4 in the serum levels of proinflammatory cytokines | From baseline visit through the safety follow-up visit on Day 43
Change from baseline through Week 4 in messenger RNA transcriptome levels on the skin. | From baseline visit through the safety follow-up visit on Day 43

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Kymera Investigative Site, Birmingham, Alabama
  - Kymera Investigative Site, Fountain Valley, California
  - Kymera Investigative Site, Santa Monica, California
  - Kymera Investigative Site, Boynton Beach, Florida
  - Kymera Investigative Site, Hollywood, Florida
  - Kymera Investigative Site, Tampa, Florida
  - Kymera Investigative Site, Fargo, North Dakota
  - Kymera Investigative Site, Dublin, Ohio
  - Kymera Investigative Site, Springfield, Ohio
  - Kymera Investigative Site, Tulsa, Oklahoma
  - Kymera Investigative Site, Charleston, South Carolina
  - Kymera Investigative Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No